CLINICAL TRIAL: NCT01055002
Title: A Pilot Phase II Study of the Efficacy of Antimalarial Drugs Against Plasmodium Falciparum by Experimental Challenge With a Low Dose of Blood Stage Parasites in Healthy Male Volunteers
Brief Title: A Pilot Study to Test Activity of Antimalarial Drugs Against an Induced Malaria Infection in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Queensland Institute of Medical Research (Other); Q-Pharm Pty Limited (Industry); Trident Clinical Research Pty Ltd (Industry)
Responsible Party: Dr James McCarthy, Queensland Institute of Medical Research
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: QP09C08
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Healthy; Non-smokers
Keywords: Health male volunteers; Male volunteers aged 18-45 years; Non-smokers and in good health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artemether/lumefantrine tablets (Active Comparator): Artemether (20 mg) and Lumefantrine (120 mg) tablets: Four tablets taken as a single dose twice a day with fatty food for three days (total dose of 24 tablets in 6 doses) on days 6-8
  Interventions: Biological: Blood stage parasite (BSP) inoculum
- Atovaquone/Proguanil HCl tablets (Active Comparator): Atovaquone (250 mg) and Proguanil HCl (100 mg) tablets: Four tablets taken as a single dose daily for 3 days (total dose of 12 tablets) on days 6-8
  Interventions: Biological: Blood stage parasite (BSP) inoculum

INTERVENTIONS:
Biological: Blood stage parasite (BSP) inoculum — Inoculum of human red blood cells infected with falciparum malaria administered intravenously on Day 1

SUMMARY:
This is a pilot study of a protocol for inducing a falciparum malaria infection in healthy volunteers in order to test the activity of novel agents being developed as drugs for the treatment of uncomplicated malaria. In this pilot study, 16 healthy male volunteers will be administered a low level malaria infection via infected human red blood cells. After 6 days they will be administered one of two registered antimalarial treatments (8 volunteers for each treatment) in order to define the rate of clearance of the infection. This information will be used to design similar future studies for the initial assessment of the efficacy of novel antimalarial drugs in development.

DETAILED DESCRIPTION:
This is a single-center, controlled, randomized, study using a BSP inoculum challenge as a model to assess the activity of antimalarial agents. The study will be conducted in 2 cohorts (n = 6 and n = 10). Cohort 2 will not commence until at least after day 12 of cohort 1 and review by Safety Review Team following day 9 exit of cohort 1. The participants will be randomized 1:1 to the two registered antimalarials. This is an enabling study using registered antimalarial drugs as reference treatments (one slow acting and one fast acting), aimed to inform trial design, endpoints and testing regimens for assessing new candidate antimalarial drugs in development. The study will follow the sequence of the challenge inoculation, reference treatment and follow-up.

Healthy male participants will be inoculated on Day 1 with ~1,800 Plasmodium falciparum-infected human erythrocytes administered intravenously. On an outpatient basis, participants will be monitored morning (AM) and night (PM) from day 3 to day 5 for adverse events and the unexpected early onset of symptoms, signs or parasitological evidence of malaria. On day 5 evening, participants will be admitted to the study unit and confined for safety monitoring and antimalarial treatment. Reference treatment administration will begin on the evening of Day 6 and continued on Day 7 and 8 (3 days of treatment).

If clinical or parasitologic evidence of malaria (either the identification of two or more malaria parasites on a malaria thick film, platelet count less than 100 x109/L, or the onset of clinical features of malaria) occurs before day 6 evening, allocated treatment will begin at this time.

Following treatment, participants will be followed up as inpatients for at least 86 hours, (4 evenings) to ensure tolerance of the therapy and clinical response, then if clinically well on an outpatient basis for safety and continued presence of malaria parasites via PCR and thick blood film review.

Adverse events will be monitored via telephone monitoring, within the clinical research unit and on outpatient review after malaria challenge inoculation and antimalarial study drug administration. Blood samples for safety evaluation, malaria monitoring, and red blood cell antibodies will be drawn at baseline and at nominated times after malaria challenge.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-45 years who do not live alone
* BMI within 18-30
* Understand the procedures and risks involved
* Contactable for the duration of the study
* Non-smokers and in good health
* Good venous access

Exclusion Criteria:

* History of malaria
* Been in a malaria-endemic country within 12 months
* Evidence of cardiovascular risk
* Splenectomy
* History of severe allergic reactions after vaccination of infusion
* Any serious chronic illness
* Inherited genetic anomaly
* Any volunteers wishing to donate blood to the blood bank in the future
* Retinal or visual field changes
* Diagnosis of chronic severe psychiatric condition
* Hospitalisation within 5 years for psychiatric illness, suicide attempt or danger to self or others
* Receiving psychiatric drugs (some exceptions)
* Known QTc prolongation
* Family history of cardiac anomalies
* Recent or current therapy with an antibiotic or drug with potential antimalarial activity
* Known hypersensitivity to artemether or lumefantrine, atovaquone or proguanil hydrochloride or any of the excipients
* Concomitant use of any drug which is metabolised by the cytochrome enzyme CYP2D6 OR drugs that are known to prolong the QTc interval
* Use of corticosteroids, anti-inflammatory drugs, any immunomodulators or anticoagulants. Currently receiving or have previously received immunosuppressive therapy, including systemic steroids including ACTH or inhaled steroids in dosages which are associated with hypothalamicpituitary- adrenal axis suppression such as 1mg/kg/day of prednisone or its equivalent or chronic use of inhaled high potency corticosteroids
* Presence of acute infectious disease or fever
* Evidence of acute illness within the four weeks before trial prior to screening
* Significant intercurrent disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmune disease by history, physical examination, and/or laboratory studies including urinalysis
* Alcohol consumption greater than community norms
* A history of drug habituation, or any prior intravenous usage of an illicit substance
* Medical requirement for intravenous immunoglobulin or blood transfusions
* Participation in any investigational product study within the 8 weeks preceding the study
* Participation in any research study involving significant blood sampling, or blood donation to a blood bank during the 8 weeks preceding the study
* Have ever received a blood transfusion
* Positive test for HIV, Hepatitis B, hepatitis C, Human T-cell Lymphotropic Virus I & II (HTLVI & HTLVII), and syphilis
* Any clinically significant biochemical or haematologic abnormality (Hb must be ≥13.5g/dL)
* Ingestion of any poppy seeds within the 48 hours prior to the screening blood test
* Detection of any recreational drug listed in the urine drug screen

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Parasite clearance rates by PCR | 1-7 days after drug treatment

SECONDARY OUTCOMES:
Parasite growth rates by PCR | 1-6 days after inoculation

CONTACTS AND LOCATIONS:
Overall Officials: James McCarthy, MD FRACP, Principal Investigator — Queensland Institute of Medical Research
Locations (1):
- Q-Pharm Clinics, Royal Brisbane and Women's Hospital, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] McCarthy JS, Sekuloski S, Griffin PM, Elliott S, Douglas N, Peatey C, Rockett R, O'Rourke P, Marquart L, Hermsen C, Duparc S, Mohrle J, Trenholme KR, Humberstone AJ. A pilot randomised trial of induced blood-stage Plasmodium falciparum infections in healthy volunteers for testing efficacy of new antimalarial drugs. PLoS One. 2011;6(8):e21914. doi: 10.1371/journal.pone.0021914. Epub 2011 Aug 22. PMID 21887214